CLINICAL TRIAL: NCT00406952
Title: A Phase 4 Randomized, Double-Blind, Placebo Controlled Methodology Study to Evaluate the Time of Onset of AntiDepressant Response in Subjects With Major Depressive Disorder
Brief Title: Study for Evaluating Different Methods of Measuring Depression Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A9001337
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

INTERVENTIONS:
Procedure: electronic diary
Drug: Sertraline
Drug: Placebo
Procedure: voice acoustics

SUMMARY:
Purpose of the study is to evaluate use of electronic diaries and voice acoustics for use in future depression clinical trial. Focus is on increased precision of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder with symptoms of depression present at least 1 month
* Psychotropic medications currently not being taken

Exclusion Criteria:

* Failure to respond in past 5 years to antidepressant therapy of adequate duration and dosing
* Diagnoses of following conditions or disorders within past 6 months: generalized anxiety, obsessive compulsive, panic, post stress, anorexia, bulimia, alcohol or substance abuse or social anxiety disorder
* Diagnoses current or past of the following conditions or disorders: schizophrenia, psychotic disorder, delieium, dememtia, amnestic cognitive disorder, bipolar

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2006-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is time to treatment response and difference in time to response for the two data collection methods - daily patient electronic assessment versus weekly assessments measured in clinic.

SECONDARY OUTCOMES:
The secondary endpoint is the difference in study participation burden between standard and enhanced data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Elmsford, New York
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Midvale, Utah

REFERENCES:
- [Derived] Mundt JC, Vogel AP, Feltner DE, Lenderking WR. Vocal acoustic biomarkers of depression severity and treatment response. Biol Psychiatry. 2012 Oct 1;72(7):580-7. doi: 10.1016/j.biopsych.2012.03.015. Epub 2012 Apr 26. PMID 22541039
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001337&StudyName=Study%20for%20evaluating%20different%20methods%20of%20measuring%20depression%20%20treatment%20response%20